CLINICAL TRIAL: NCT03819712
Title: Identification of Predictive Blood Biomarkers of Recurrent Urinary Tract Infections
Acronym: Predict-UTI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 18-PP-05
Record Dates: First submitted 2019-01-25; First posted 2019-01-28 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Urinary Tract Infections
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No recurrent UTI (Experimental): Healthy female volunteer aged 18 to 28 years reporting a single cystitis since the age of 14 years
  Interventions: Procedure: Collection of blood samples; Other: Collection of fecal samples; Other: Collection of urine samples; Other: Collection of vaginal swaps
- Recurrent UTI (Experimental)
  Interventions: Procedure: Collection of blood samples; Other: Collection of fecal samples; Other: Collection of urine samples; Other: Collection of vaginal swaps

INTERVENTIONS:
Procedure: Collection of blood samples — 23 mL of blood will be collected during the inclusion visit
Other: Collection of fecal samples — Fecal sample self-collected after the inclusion visit
Other: Collection of urine samples — 10 mL of urine will be collected during the inclusion visit
Other: Collection of vaginal swaps — Sample of vaginal microbiota collected during the inclusion visit

SUMMARY:
Urinary tract infections affect more than 130 million people worldwide each year. Almost 50% of women will have at least one urinary tract infection during their lifetime, usually cystitis. Half of them will have recurrent cystitis. Antibiotics are the first-line treatment for cystitis, but their effectiveness is decreasing due to the rapid spread of multi-resistant uro-pathogenic bacteria. The objective of this study is to identify blood biomarkers associated with a high risk of recurrent cystitis. Immune system cells, and more specifically innate immunity cells, play a key role in controlling urinary tract infections. In addition, clinical studies have shown that there is a high inter-individual variability in the ability of innate immune cells to respond to different stimuli. We therefore hypothesized that there was an association between the risk of recurrent cystitis and a deficiency of certain immune cell types in producing certain pro-inflammatory cytokines, including TNF-α, in response to one or more bacterial stimuli, particularly flagellin.

ELIGIBILITY:
Inclusion Criteria:

* Female aged 18 to 28 years;
* Subject accepting to be serologically tested for HIV and HCV;
* Subject considered healthy by the physician on the basis of medical history and clinical examination;
* Subject with a body mass index between 18.5 and 30 kg/m2;
* Subject understands and speaks French and is able to give written consent;
* Subject affiliated to Social Security or a similar regime;
* Having reported a single cystitis since the age of 14 (Group 1), or 3 or more cystitis over a 12-month period since the age of 14 (Group 2).

Exclusion Criteria:

* Subject protected by law under guardianship or curatorship, or unable to participate in a clinical study under Article L. 1121-16 of the French Public Health Code;
* Subject who has participated in a clinical research study in the last 3 months in which he/she was exposed to a pharmaceutical product or medical device;
* Subject who has stayed in a tropical or subtropical country in the last 3 months;
* Pregnant or breastfeeding subject for women of childbearing age;
* Subject with special diet for medical reasons and prescribed by a doctor or dietician (e.g. a low-calorie diet or a diet intended to lower cholesterol levels);
* Subject who regularly consumes large quantities of alcohol, i. e. more than 50 g of pure alcohol per day (e. g. more than 4 glasses of 150 ml wine, more than 4 pints of 250 ml beer, or more than 4 glasses of 40 ml containing strong alcohol);
* Subject who has used an illegal recreational drug in the past 3 months;
* Subject who has taken an immunosuppressive or immunomodulatory drug (excluding intranasally or topically administered corticosteroids) in the past 2 weeks, or for more than 14 consecutive days in the past 6 months;
* Subject who has been vaccinated within the last 3 months;
* Subject who received a blood transfusion or immunoglobulins in the last 3 months;
* Subject stating that he has not been fasting for at least 10 hours;
* Subject reporting HIV or HCV status;
* Subject who had an infectious episode or was treated with antibiotics during the 4 weeks prior to the visit;
* Subject with a positive urinary pregnancy test;
* Subject with a severe and/or chronic and/or recurrent pathology, in particular:

  * A chronic inflammatory and/or autoimmune or allergic disease and in particular a chronic inflammatory disease of the intestine (Crohn's disease, ulcerative colitis), epidermis (psoriasis, atopic dermatitis), joints (rheumatoid arthritis), nervous system (multiple sclerosis), type I diabetes;
  * High blood pressure or type II diabetes;
  * A neurodegenerative disease.
* Subject who has been diagnosed with cancer and has not been in remission for more than 5 years.

Ages: 18 Years to 28 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 109 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2023-12-03 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
TNF-α measurement in blood cell culture media using Luminex® technology. | At 18 months
  The concentrations of TNF-α will be expressed in ng/ml by calibration with a standard range.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital de l'Archet 1 - CHU de Nice - Service d'Infectiologie, Nice, France

IPD SHARING:
Plan to Share IPD: Undecided